CLINICAL TRIAL: NCT02520011
Title: Phase 2, Randomized, Biomarker-driven Clinical Study in Patients With Relapsed or Refractory Acute Myeloid Leukemia (AML) With MCL-1 Dependence ≥30%
Brief Title: Alvocidib Biomarker-driven Phase 2 AML Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow enrollment, the extensive time projected to conclude the study hypothesis rendered the study no longer reasonably feasible to complete.
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TPI-ALV-201
Record Dates: First submitted 2015-08-06; First posted 2015-08-11 (Estimated); Results first posted 2021-07-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Acute Myeloid Leukemia
Keywords: Refractory AML; Relapsed AML; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — alvocidib; Cytarabine; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ACM (Stage 1 / Stage 2) (Experimental): A: alvocidib, 30 mg/m2 as a 30 minute intravenous (IV) bolus followed by 60 mg/m2 over 4 hours as an IV infusion administered daily on Days 1-3; C: cytarabine (ara-c), 2 gm/m2 by continuous IV infusion over 72 hours on Days 6-8; M: mitoxantrone (mitoxantrone hydrochloride), 40 mg/m2 by IV infusion over 1-2 hours starting 12 hours after completing cytarabine
  Interventions: Drug: Alvocidib; Drug: Cytarabine; Drug: Mitoxantrone
- CM (Stage 2) (Active Comparator): C: cytarabine (ara-c), 2 gm/m2 by continuous IV infusion over 72 hours on Days 1-3; M: mitoxantrone (mitoxantrone hydrochloride), 40 mg/m2 by IV infusion over 1-2 hours starting 12 hours after completing cytarabine
  Interventions: Drug: Cytarabine; Drug: Mitoxantrone

INTERVENTIONS:
Drug: Alvocidib
  Arms: ACM (Stage 1 / Stage 2)
Drug: Cytarabine
  Other Names: ara-c
Drug: Mitoxantrone
  Other Names: mitoxantrone hydrochloride

SUMMARY:
The purpose of this two-stage Phase 2 study is to assess the clinical response (Complete Remission) of ACM (Alvocidib/Cytarabine/Mitoxantrone) compared to CM (Cytarabine/Mitoxantrone) treatment in refractory or relapsed AML patients with demonstrated MCL-1 dependence of ≥ 30% by mitochondrial profiling in bone marrow.

DETAILED DESCRIPTION:
In Stage 1 of the study, all eligible AML patients with demonstrated MCL-1 dependence of ≥ 30% by mitochondrial profiling in bone marrow will receive treatment with ACM.

In Stage 2, all eligible AML patients with demonstrated MCL-1 dependence of ≥ 30% by mitochondrial profiling in bone marrow will be randomized 1:1 to receive either treatment with ACM or CM.

ELIGIBILITY:
Inclusion Criteria:

1. Be between the ages of ≥18 and ≤65 years
2. Have an established, pathologically confirmed diagnoses of AML by World Health Organization (WHO) criteria excluding acute promyelocytic leukemia (APL-M3) with a bone marrow of >5% blasts based on histology or flow cytometry
3. Be in first relapse (within 24 months of CR) or have failed induction therapy* (no CR or CRi after treatment with an intensive regimen (eg, anthracycline/cytarabine ± etoposide, gemtuzumab ozogamicin, or cladribine).

   *Induction therapy may involve 1 or 2 cycles of the same regimen. Efficacy assessment of induction therapy must be >21 days from the start of the previous induction cycle.
4. Demonstrate MCL-1 dependence of ≥30% by mitochondrial profiling in bone marrow.
5. Have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤2
6. Have a serum creatinine level ≤1.8 mg/dL
7. Have an alanine aminotransferase (ALT)/aspartate aminotransferase (AST) level ≤5 times upper limit of normal (ULN)
8. Have a total bilirubin level ≤2.0 mg/dL (unless secondary to Gilbert syndrome, hemolysis, or leukemia)
9. Have a left ventricular ejection fraction (LVEF) >45% by echocardiogram (ECHO) or multigated acquisition (MUGA) scan
10. Be nonfertile or agree to use an adequate method of contraception. Sexually active patients and their partners must use an effective method of contraception associated with a low failure rate during and for at least 6 months after completion of study therapy.
11. Be able to comply with the requirements of the entire study.
12. Provide written informed consent prior to any study related procedure.

Exclusion Criteria:

1. Received more than 2 cycles of induction therapy for AML. Investigational agents as part of front-line therapy for AML may by acceptable following discussion with the Medical Monitor. Hydroxyurea is permitted (see #5 below).
2. Received any previous treatment with alvocidib or any other CDK inhibitor
3. Received a hematopoietic stem cell transplant within the previous 2 months
4. Have clinically significant graft versus host disease (GVHD), or GVHD requiring initiation or escalation of treatment within the last 21 days
5. Require concomitant chemotherapy, radiation therapy, or immunotherapy. Hydroxyurea is allowed up to the evening before starting (but not within 12 hours) of starting treatment on either arm.
6. Received >360 mg/m2 equivalents of daunorubicin
7. Have a peripheral blast count of >30,000/mm3 (may use hydroxyurea as in #5 above)
8. Received antileukemic therapy within the last 3 weeks (with the exception of hydroxyurea or if the patient has definite refractory disease). Refractory patients who received therapy within the last 3 weeks may be eligible with prior approval of the Medical Monitor.
9. Diagnosed with acute promyelocytic leukemia (APL, M3)
10. Have active central nervous system (CNS) leukemia
11. Have evidence of uncontrolled disseminated intravascular coagulation
12. Have an active, uncontrolled infection
13. Have other life-threatening illness
14. Have other active malignancies or diagnosed with other malignancies within the last 6 months, except nonmelanoma skin cancer or cervical intraepithelial neoplasia
15. Have mental deficits and/or psychiatric history that may compromise the ability to give written informed consent or to comply with the study protocol.
16. Are pregnant and/or nursing
17. Have received any live vaccine within 14 days prior to first study drug administration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2016-03-14 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Anthony, DO, Study Director — Sumitomo Pharma America, Inc.
Locations (38):
- United States (26):
  - Honor Health Research Institute, Scottsdale, Arizona
  - University of California Los Angeles (UCLA), Los Angeles, California
  - University of California San Diego UCSD, San Diego, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - Northside Hospital, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Westwood, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Sidney Kimmel Cancer Center at Johns Hopkins, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Morristown Cancer Center, Morristown, New Jersey
  - Roswell Park Cancer Center Institute, Buffalo, New York
  - Hudson Valley Cancer Center, Hawthorne, New York
  - Columbia University Medical Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - West Penn Allegheny Hospital, Pittsburgh, Pennsylvania
  - Baylor Sammons Cancer Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Princess Margaret Cancer Center, Toronto, Ontario, Canada
- Spain (8):
  - Hospital Regional Universitario de Malaga, Málaga, Malaga
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Institut Catala d'Oncologia, Badalona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Universitario Central de Asturias - HUCA, Oviedo
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitari i Politècnic La Fe, Valencia
- United Kingdom (3):
  - University Hospitals of Wales, Cardiff, Wales
  - Univ Hospital of Bristol, Bristol
  - Guys Hospital St. Thomas, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolled 104 pts from 14Mar2016 to 12Feb2020 at 22 of 40 sites. Patients were hospitalized until completion of their chemotherapy. The study terminated early in Jan2020 due to a steady and marked reduction in enrollment. The study protocol underwent a few major amendments during the course of the trial. Although the study protocol and the SAP had planned for comprehensive analysis of the efficacy data, only select efficacy analyses could be performed due to early termination of the trial.
Groups:
- CM Relapsed/Refractory: Patients who were relapsed/refractory AML and were enrolled during Stage 2 and received Cytarabine 2 gm/m2 by continuous infusion over 72 hours on Days 1-3 and Mitoxantrone 40 mg/m2 by IV over 1-2 hours starting 12 hours after completing cytarabine.
- ACM Relapsed/Refractory: Patients who had relapsed/refractory AML and were enrolled during Stage 1 and Stage 2 and received Alvocidib 30 mg/m2 as a 30-minute intravenous bolus followed by 60 mg/m2 over 4 hours as an IV infusion administered daily on Days 1-3 with Cytarabine 2 gm/m2 by continuous IV infusion on Days 6-8 and Mitoxantrone 40 mg/m2 by IV infusion over 1-2 hours starting 12 hours after completing cytarabine.
- ACM Newly Diagnosed: Patients who were newly diagnosed AML and enrolled during Stage 1 and Stage 2 and received Alvocidib 30 mg/m2 as a 30-minute intravenous bolus followed by 60 mg/m2 over 4 hours as an IV infusion administered daily on Days 1-3 with Cytarabine 2 gm/m2 by continuous IV infusion on Days 6-8 and Mitoxantrone 40 mg/m2 by IV infusion over 1-2 hours starting 12 hours after completing cytarabine.
Period: Overall Study
Arm/Group | CM Relapsed/Refractory | ACM Relapsed/Refractory | ACM Newly Diagnosed
Started | 11 | 79 | 14
Stage 1 | 0 | 32 | 10
Stage 2 | 11 | 47 | 4
Completed | 6 | 33 | 5
Not Completed | 5 | 46 | 9
Not completed — Adverse Event | 0 | 1 | 2
Not completed — Death | 0 | 8 | 1
Not completed — Lack of Efficacy | 4 | 26 | 4
Not completed — Physician Decision | 0 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 0
Not completed — Protocol Deviation | 0 | 1 | 0
Not completed — Patient went to hospice | 0 | 1 | 0
Not completed — Progressive disease following response | 0 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- CM Relapsed/Refractory: Stage 2 Relapsed/Refractory AML patients who were randomized to receive CM
- ACM Relapsed/Refractory: Relapsed/Refractory AML patients enrolled to Stage 1 and those enrolled to Stage 2 who received ACM.
- ACM Newly Diagnosed: Newly diagnosed AML patients enrolled and received ACM.
- Total: Total of all reporting groups
Arm/Group | CM Relapsed/Refractory | ACM Relapsed/Refractory | ACM Newly Diagnosed | Total
Number analyzed (Participants) | 11 | 79 | 14 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 79 | 14 | 104
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 40 | 3 | 47
  Male | 7 | 39 | 11 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 4 | 0 | 4
  White | 11 | 70 | 13 | 94
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 1 | 4
2017 ELN genetic risk criteria classification [Count of Participants; unit: Participants] — Per the 2017 ELN genetic risk criteria, patients were classified as having an adverse, intermediate, or favorable genetic risk.
  Participants
    Adverse | 8 | 26 | 3 | 37
    Intermediate | 1 | 13 | 0 | 14
    Favorable | 2 | 6 | 1 | 9
    Missing | 0 | 34 | 10 | 44

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) Rate in Patients With Relapsed or Refractory AML
Description: Complete Remission (CR) rate = Percentage of patients achieving CR after Cycle 1 as defined in Stage 1 by the International Working Group (IWG) Criteria and 2010 European LeukemiaNet (EN) criteria in patients with relapsed or refractory AML with MCL-1 dependence >30% and in Stage 2 by the 2017 ELN criteria.
  The study was terminated in January 2020 due to a steady and marked reduction in enrollment. Thus, the efficacy endpoints could not be analyzed. As sufficient efficacy results were not available to analyze patients based on the percentage of MCL-1 dependency the treatment efficacy was summarized by distributing the safety population into 6 groups based on whether the patients received the ACM vs CM regimen and their disease stages at study entry.
Time Frame: Best response after at least 1 cycle through study completion approximately 4 years
Measure: Number; unit: participants
Groups:
- Stage 2 CM Relapsed/Refractory: Stage 2 Relapsed/Refractory AML patients who were randomized to receive CM
- Stage 2 ACM Relapsed/Refractory: Stage 2 Relapsed/Refractory AML patients who were randomized to receive ACM
- Stage 1 ACM Relapsed/Refractory: Stage 1 Relapsed/Refractory AML patients received ACM
- Stages 1 and 2 ACM Relapsed/Refractory: Stages 1 and 2 Relapsed/Refractory AML patients combined who received ACM
- Stage 1 Newly Diagnosed ACM: Stage 1 Newly Diagnosed AML patients who received ACM
- All Stages and Cohorts (Including Randomized Stage): ACM Total: Total patients who received ACM (Stages 1 and 2 Relapsed/Refractory AML patients and Newly Diagnosed patients combined)"
Arm/Group | Stage 2 CM Relapsed/Refractory | Stage 2 ACM Relapsed/Refractory | Stage 1 ACM Relapsed/Refractory | Stages 1 and 2 ACM Relapsed/Refractory | Stage 1 Newly Diagnosed ACM | All Stages and Cohorts (Including Randomized Stage): ACM Total
Number analyzed (Participants) | 11 | 11 | 25 | 79 | 14 | 93
participants
  Complete Remission (CR) | 6 | 2 | 8 | 21 | 6 | 27
  CR with Incomplete Neutrophil Recovery (Cri) | 0 | 3 | 5 | 15 | 2 | 17
  Partial Remission (PR) | 0 | 0 | 1 | 1 | 1 | 2
  Resistant/Relapsed Disease | 5 | 5 | 5 | 30 | 4 | 34
  Not Evaluated | 0 | 1 | 6 | 12 | 1 | 13

2. Other Pre Specified Outcome: Response to Treatment
Description: To determine if treatment with ACM can induce CR in patients with relapsed or refractory AML with MCL-1 dependence of >30% who failed to achieve CR following 1 cycle of CM
Time Frame: Best response after at least 1 cycle through study completion approximately 4 years
Population: A total 11 patients were initially randomized to the CM arm. 6 had CR from receiving CM so they did not cross over to receive ACM. Of the remaining 5 patients, only 2 crossed over to receive ACM and were included in the analysis of this outcome.
Measure: Number; unit: participants
Groups:
- Stage 2 CM Relapsed/Refractory AML: A total 11 patients were initially randomized to the CM arm. 6 had CR from receiving CM so they did not cross over to receive ACM. Of the remaining 5 patients, only 2 crossed over to receive ACM and were included in the analysis of this outcome.
Arm/Group | Stage 2 CM Relapsed/Refractory AML
Number analyzed (Participants) | 2
participants
  Partial Remission (PR) | 1
  Not Evaluated | 1

ADVERSE EVENTS:
Time Frame: Beginning at 1st dose of study drug through 30 days of the last administration of study drug, up to 4 years.
Groups:
- CM Relapsed/Refractory: CM Relapse/Refractory patients who received at least 1 dose of study drug
- ACM Relapsed/Refractory: ACM Relapsed/Refractory patients who received at least 1 dose of study drug
- ACM Newly Diagnosed: ACM Newly Diagnosed patients who received at least 1 dose of study drug
- ACM Total: ACM Total patients who received at least 1 dose of study drug
Arm/Group | CM Relapsed/Refractory | ACM Relapsed/Refractory | ACM Newly Diagnosed | ACM Total
All-Cause Mortality (participants affected / at risk) | 1/11 | 11/79 | 1/14 | 12/93
Serious Adverse Events (participants affected / at risk) | 3/11 | 31/79 | 4/14 | 35/93
Other Adverse Events (participants affected / at risk) | 11/11 | 79/79 | 14/14 | 93/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CM Relapsed/Refractory (N=11) | ACM Relapsed/Refractory (N=79) | ACM Newly Diagnosed (N=14) | ACM Total (N=93)
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Disease progression (General disorders) | 0 | 2 | 0 | 2
Liver injury (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 3 | 1 | 4
Sepsis (Infections and infestations) | 2 | 11 | 1 | 12
Lung infection (Infections and infestations) | 0 | 3 | 1 | 4
Bacteraemia (Infections and infestations) | 0 | 2 | 0 | 2
Septic shock (Infections and infestations) | 0 | 2 | 0 | 2
Abscess neck (Infections and infestations) | 0 | 1 | 0 | 1
Anorectal infection (Infections and infestations) | 0 | 1 | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Device related infection (Infections and infestations) | 0 | 1 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1 | 0 | 1
Enterocolitis viral (Infections and infestations) | 0 | 1 | 0 | 1
Klebsiella sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia fungal (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 1 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 3 | 0 | 3
Syncope (Nervous system disorders) | 0 | 1 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CM Relapsed/Refractory (N=11) | ACM Relapsed/Refractory (N=79) | ACM Newly Diagnosed (N=14) | ACM Total (N=93)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 42 | 6 | 48
Anaemia (Blood and lymphatic system disorders) | 2 | 25 | 2 | 27
Leukopenia (Blood and lymphatic system disorders) | 0 | 7 | 5 | 12
Neutropenia (Blood and lymphatic system disorders) | 0 | 7 | 1 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 6 | 2 | 8
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 4
Splenic haematoma (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 9 | 4 | 13
Tachycardia (Cardiac disorders) | 0 | 7 | 2 | 9
Sinus bradycardia (Cardiac disorders) | 0 | 3 | 2 | 5
Atrial fibrillation (Cardiac disorders) | 0 | 4 | 0 | 4
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 2 | 2
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 2 | 2 | 0 | 2
Mydriasis (Eye disorders) | 0 | 0 | 1 | 1
Ocular discomfort (Eye disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 66 | 11 | 77
Nausea (Gastrointestinal disorders) | 8 | 44 | 9 | 53
Vomiting (Gastrointestinal disorders) | 2 | 31 | 7 | 38
Abdominal pain (Gastrointestinal disorders) | 1 | 22 | 6 | 28
Constipation (Gastrointestinal disorders) | 4 | 16 | 5 | 21
Stomatitis (Gastrointestinal disorders) | 0 | 14 | 3 | 17
Dry mouth (Gastrointestinal disorders) | 2 | 10 | 1 | 11
Haemorrhoids (Gastrointestinal disorders) | 1 | 5 | 3 | 8
Abdominal distension (Gastrointestinal disorders) | 1 | 7 | 0 | 7
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 6 | 1 | 7
Colitis (Gastrointestinal disorders) | 1 | 4 | 2 | 6
Proctalgia (Gastrointestinal disorders) | 1 | 5 | 1 | 6
Abdominal pain upper (Gastrointestinal disorders) | 1 | 5 | 0 | 5
Dyspepsia (Gastrointestinal disorders) | 0 | 4 | 1 | 5
Ileus (Gastrointestinal disorders) | 0 | 4 | 0 | 4
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 2 | 4
Oral disorder (Gastrointestinal disorders) | 1 | 3 | 0 | 3
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 2
Gingival bleeding (Gastrointestinal disorders) | 1 | 2 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Salivary gland disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 29 | 7 | 36
Pyrexia (General disorders) | 1 | 31 | 5 | 36
Fatigue (General disorders) | 1 | 29 | 5 | 34
Chills (General disorders) | 1 | 10 | 4 | 14
Mucosal inflammation (General disorders) | 1 | 9 | 0 | 9
Chest pain (General disorders) | 0 | 5 | 0 | 5
Malaise (General disorders) | 0 | 3 | 1 | 4
Non-cardiac chest pain (General disorders) | 1 | 4 | 0 | 4
Oedema (General disorders) | 1 | 4 | 0 | 4
Pain (General disorders) | 0 | 4 | 0 | 4
Face oedema (General disorders) | 0 | 2 | 1 | 3
Disease progression (General disorders) | 1 | 2 | 0 | 2
Generalised oedema (General disorders) | 0 | 1 | 1 | 2
Drug withdrawal syndrome (General disorders) | 0 | 0 | 1 | 1
Facial pain (General disorders) | 0 | 0 | 1 | 1
Asthenia (General disorders) | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 4 | 1 | 5
Cytokine release syndrome (Immune system disorders) | 0 | 4 | 1 | 5
Graft versus host disease (Immune system disorders) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 2 | 13 | 3 | 16
Lung infection (Infections and infestations) | 1 | 6 | 3 | 8
Pneumonia (Infections and infestations) | 1 | 6 | 2 | 8
Device related infection (Infections and infestations) | 0 | 5 | 1 | 6
Sinusitis (Infections and infestations) | 0 | 6 | 0 | 6
Enterococcal infection (Infections and infestations) | 0 | 5 | 0 | 5
Respiratory syncytial virus infection (Infections and infestations) | 0 | 5 | 0 | 5
Staphylococcal bacteraemia (Infections and infestations) | 0 | 5 | 0 | 5
Bacteraemia (Infections and infestations) | 0 | 4 | 0 | 4
Clostridium difficile colitis (Infections and infestations) | 0 | 4 | 0 | 4
Folliculitis (Infections and infestations) | 0 | 4 | 0 | 4
Oral herpes (Infections and infestations) | 1 | 3 | 1 | 4
Anorectal infection (Infections and infestations) | 0 | 1 | 2 | 3
Urinary tract infection (Infections and infestations) | 1 | 2 | 0 | 2
Cystitis (Infections and infestations) | 0 | 0 | 1 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 1 | 0 | 1
Enterobacter bacteraemia (Infections and infestations) | 0 | 0 | 1 | 1
Gastroenteritis Escherichia coli (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia legionella (Infections and infestations) | 0 | 0 | 1 | 1
Bronchiolitis (Infections and infestations) | 1 | 0 | 0 | 0
Groin abscess (Infections and infestations) | 1 | 0 | 0 | 0
Herpes virus infection (Infections and infestations) | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 8 | 5 | 13
Contusion (Injury, poisoning and procedural complications) | 0 | 6 | 1 | 7
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 5 | 2 | 7
Procedural pain (Injury, poisoning and procedural complications) | 0 | 4 | 0 | 4
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 3
Incision site erythema (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
White blood cell count decreased (Investigations) | 1 | 27 | 4 | 31
Alanine aminotransferase increased (Investigations) | 1 | 19 | 4 | 23
Platelet count decreased (Investigations) | 1 | 18 | 4 | 22
Aspartate aminotransferase increased (Investigations) | 1 | 19 | 2 | 21
Lymphocyte count decreased (Investigations) | 2 | 13 | 4 | 17
Neutrophil count decreased (Investigations) | 0 | 12 | 1 | 13
Weight decreased (Investigations) | 0 | 8 | 3 | 11
Blood bilirubin increased (Investigations) | 2 | 6 | 3 | 9
Blood creatinine increased (Investigations) | 0 | 6 | 0 | 6
International normalised ratio increased (Investigations) | 0 | 6 | 0 | 6
Blood lactate dehydrogenase increased (Investigations) | 0 | 4 | 1 | 5
Blood phosphorus increased (Investigations) | 0 | 4 | 1 | 5
Electrocardiogram QT prolonged (Investigations) | 0 | 4 | 1 | 5
Blood alkaline phosphatase increased (Investigations) | 0 | 4 | 0 | 4
Blood phosphorus decreased (Investigations) | 0 | 1 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 40 | 7 | 47
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 28 | 5 | 33
Decreased appetite (Metabolism and nutrition disorders) | 1 | 21 | 3 | 24
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 20 | 4 | 24
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 14 | 8 | 22
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 18 | 3 | 21
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 13 | 4 | 17
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 12 | 3 | 15
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 9 | 0 | 9
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 7 | 1 | 8
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 5 | 2 | 7
Fluid overload (Metabolism and nutrition disorders) | 1 | 6 | 0 | 6
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 15 | 1 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 1 | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 5 | 1 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 21 | 2 | 23
Dysgeusia (Nervous system disorders) | 1 | 8 | 3 | 11
Dizziness (Nervous system disorders) | 1 | 8 | 2 | 10
Syncope (Nervous system disorders) | 1 | 3 | 1 | 4
Somnolence (Nervous system disorders) | 0 | 1 | 1 | 2
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 14 | 3 | 17
Anxiety (Psychiatric disorders) | 0 | 6 | 2 | 8
Depression (Psychiatric disorders) | 1 | 6 | 0 | 6
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 1 | 1
Hallucination (Psychiatric disorders) | 1 | 1 | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 11 | 2 | 13
Haematuria (Renal and urinary disorders) | 0 | 6 | 0 | 6
Urinary retention (Renal and urinary disorders) | 0 | 2 | 1 | 3
Dysuria (Renal and urinary disorders) | 0 | 1 | 1 | 2
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 2 | 0 | 2
Acquired phimosis (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 16 | 2 | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 10 | 3 | 13
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 10 | 1 | 11
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 2 | 7
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 1 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 2 | 6
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 4
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 10 | 5 | 15
Rash (Skin and subcutaneous tissue disorders) | 1 | 13 | 1 | 14
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 9 | 2 | 11
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 5 | 1 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 6 | 0 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 4
Erythema (Skin and subcutaneous tissue disorders) | 0 | 4 | 0 | 4
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 3
Purpura (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 3
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 2 | 17 | 5 | 22
Hypertension (Vascular disorders) | 0 | 9 | 0 | 9
Orthostatic hypotension (Vascular disorders) | 0 | 4 | 1 | 5
Hot flush (Vascular disorders) | 0 | 1 | 1 | 2
Embolism (Vascular disorders) | 0 | 0 | 1 | 1

LIMITATIONS AND CAVEATS:
The protocol underwent a few major amendments to shorten time to complete and allow for an expeditious analysis and reporting of outcomes. The study was terminated early Jan 2020 due to marked decrease in enrollment and thus could not reach all of its efficacy endpoints. Only select analyses could be performed. Treatment efficacy was summarized by distributing the safety population into 6 groups based on whether the patients received ACM or CM regimen and their disease stages at study entry.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT02520011/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/11/NCT02520011/SAP_001.pdf